CLINICAL TRIAL: NCT05265442
Title: DUNE - A Real-life Observational Study of Cancer Pain Management With Methadone (Zoryon®) in Patients Inadequately Relieved by Other Level 3 Opioids.
Brief Title: Real-life Observational Study of Cancer Pain Management With Methadone
Acronym: DUNE
Status: Completed | Type: Observational
Sponsor: RECORDATI GROUP (Industry)
Responsible Party: Sponsor
Other Study IDs: METHADONE-LBR-NI-0571
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-08

CONDITIONS: Cancer Pain
MeSH Terms: conditions — Cancer Pain | interventions — Methadone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Methadone — titration of Zoryon (methadone): increase of posology untill pain relieved is reached

SUMMARY:
Study rational. Methadone is a distinctive opioid because of its pharmacological characteristics and its multiple modes of action, reinforcing its therapeutic value in managing advanced cancer pain, particularly in cases with a neuropathic component. However, the complex pharmacodynamics of methadone makes its prescription sometimes challenging. There is a wide inter-individual variability of its half-life. This long half-life is a valued characteristic for the management of patients treated for an addictive disorder. However, in the context of pain management, it greatly complicates the switch from and to another opioid, accentuating the risk of overdose. This is the reason why LBR, willing to improve his knowledge about Methadone in real life clinical practice wants to performe this study.

We anticipate that most patients will receive one of the above-described protocols, but we must anticipate that other protocols may be used in clinical practice in the absence of specific recommendations. Therefore it is of utmost relevance to describe the safety when initiating treatment with Zoryon® during the crucial period from D1 until the day of optimal dosage is determined (DOD) as the clinical practice may vary from a practician to another, and then until the routine follow-up visit one month after initiation of the treatment (D28).

DETAILED DESCRIPTION:
To describe the occurrence of overdose and QTc prolongation in patients initiating a treatment with Zoryon® for intractable cancer pain not adequately relieved from other level 3 opioids, from the day of instauration (D1) to the day of determination of the optimal dose for the patient (DOD: Day of Optimal Dosage (DOD): the dosage of Zoryon® will be considered optimal after two consecutive days without modification to the posology (usually within the first week) AND pain relief for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients with intractable cancer pain inadequately relieved by other opioids (ineffective and/or excessive adverse events) AND for whom switching from opioid to Zoryon® has been prescribed.
* be aged 15 years or older;
* suffer from cancer pain;
* be treated with a level 3 opioid with inadequate pain relief, i.e., ineffective, excessive adverse effects, or both;
* have a prescription to initiate Zoryon® treatment.

Exclusion Criteria:

* patients participating, or having participated within the previous month, in a clinical trial evaluating a new pain management treatment will be excluded, except for patients participating in the French experimentation of the use of therapeutical cannabis

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with intractable cancer pain inadequately relieved by other opioids (ineffective and/or excessive adverse events) AND for whom switching from opioid to Zoryon® has been prescribed.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of patients suffering from either one or the other following complications from D1 to DOD | around one week
  * Overdose episode, defined by a Richmond score ≤ -4 and a respiratory rate < 8 / min
  * QTc prolongation episode, defined by an episode > 500 ms (grade 3 according to CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Gisele Chvetzoff, Pr, Principal Investigator — CLCC Leon Berard- Lyon - France
Locations (1):
- LBR, Puteaux, France

IPD SHARING:
Plan to Share IPD: No